CLINICAL TRIAL: NCT02992587
Title: Frailty In Cardiac Surgery Copenhagen Study
Acronym: FICS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christian Holdflod Møller, Doctor of Medical Science, Rigshospitalet, Denmark
Other Study IDs: H-15004343
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Comprehensive Assessment of Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: CAF, Comprehensive assessment of frailty — CAF, Comprehensive assessment of frailty. A scoring system of the patients physical status. By smaller physical test of balance, strength and walking speed.

SUMMARY:
Background:

Over the past decades there have been seen an increase in life expectancy in Denmark. One of the consequences is that the patients who need heart surgery have a higher average age and some of these patients have a fragile physique that increases the risks of major surgery.

In cardiac surgery, there are different types of scoring system for assessing the preoperative risk of death associated with surgery. Among them are EuroSCORE and STS systems the most used.

This study evaluate the preoperative risk using the frailty score system, CAF (comprehensive assessment of frailty), based on an assessment of the patient's physical condition. If the patient has a lower than expected physical condition, the patient is frail. The assessment of the physical condition generated from questions about the patient's medical history and physical activity as well as performing less physical tests, consisting of strength, balance and walking speed.

Purpose:

A prospective observational study, who investigates how many of the patients who must undergo heart surgery, that is frail. Then compare the patients who are frail with non-frail patients in terms of complications, mortality and quality of life after the procedure. By use of CAF score the patients are scored frail or non-frail. There is planned a further study which compare degree of kidney injury in frail with non-frail patients. Our assumption is that patients which are frail, have an increased risk of complications and longer hospital stay, higher consumption of intensive days and more readmissions. Using frailty score in combination with the existing score systems EuroSCORE and STS score, are believed to be a better predictor of complications following heart surgery.

Method:

FICS study is a prospective observational study of patients undergoing cardiac surgery in the cardiothoracic department of Rigshospitalet. Planned to enroll 600 patients over a two year period. The study consists of various smaller physical test and questions. Which is used to assess whether the patient is frail and not frail.

Postoperatively follow-up after 30 days with a phone call and after 12 months through danish data register. At the both follow-up times, data are collected on the somatic readmissions / diagnoses and vital status through the national register and review of relevant journal notes. Afterwards comparing complications and mortality.

Who can enter:

One patients can be included if the following criteria are met: Age> 65 years, Elective or subacute surgery, CABG (coronary artery bypass grafting),valve substitution or combination of these

If one or more of the following criteria are met, the patient is not included in the study:

Acute surgery, Clinical unstable, Severe neuropsychiatric impairment, Uncooperative (psychiatric diagnosis) and Re-operations.

Side effects, risks and disadvantages:

Today preoperative risk assessment are assessed by EuroSCORE. Introduction of CAF, frailty score will not expose patients to the risk or side effect, since the course or treatment does not change.

Economy:

There are considered that the study are economically justified, since hypothetically this would lead to fewer readmissions, fewer days in intensive care and shorter hospital.

Acquisition:

The patients will in this trial be over 65 years old and must have completed elective or subacute cardiac surgery. They will receive participant information and thus the opportunity to read about the study before the first appearance.

At first appearance they meet our project assistant and get here verbal information about the study, where also questions can be answered. Subsequently, the patients will be asked to sign a consent form.

Publication of test results / research ethics statement:

The knowledge and results obtained through the survey will provide essential scientific information of significance for the future course and treatment of patients undergoing cardiac surgery with regard to the number of hospital days, intensive days and readmissions. Thus, the investigator believes that the study is appropriate and ethically

DETAILED DESCRIPTION:
Background:

In general, patients referred to cardiac surgery are aging. An increasing number of patients are now older than 70 years. [1]This older population of patients undergoing cardiac surgery often has several comorbidities and has an increased risk of complications and mortality compared to the younger patients.[1,2] Furthermore, several studies have shown that elderly patients with cardiovascular diseases may be frail. Frailty is a term used to assess the true biological status of a patient and defined as a patient's impaired resistance to stressors due to a decline in physiologic reserve.[3-8] In cardiac surgery there are several risk scores to assess 30-day mortality exists. The most common are the European system for cardiac operative risk evaluation (EuroSCORE) I, EuroSCORE II and the Society of Thoracic Surgeons (STS) score. However, the EuroSCORE seems to have a tendency to overestimate the perioperative risk in the elderly population and opposite the STS score a tendency to underestimate the risk. One of the reasons for this may be that none of the risk scores incorporate the biological status of the patients.[9-11] Within the last 5 years a few studies evaluating different 'frailty scores' in cardiac patients has been published. [3-6,8,12-16] None of these frailty risk scores are fully validated and therefore widely adopted. In a German single center study of 400 patients undergoing elective cardiac surgery and aged 74 or above frailty was assessed by the comprehensive assessment of frailty (CAF) score. The CAF scores assess weakness, self-reported exhaustion, slowness of gait speed, low activity and physical performance. [14,15] The CAF score correlates well with the EuroSCORE and STS score, but is a very complex and time consuming risk score. In an effort to make the test more clinical practical a simpler version of the CAF score has been developed. The 'frailty predicts death one year after elective cardiac surgery test' (FORECAST) includes; chair rise, self-reported weakness, stair climbing, two physicians estimation of frailty and serum creatinine level. [14,17]

Aim:

In an observational prospective study, we will identify and describe the number of frail patients undergoing first time cardiac surgery in our department, compare the risk of short-term and long-term complications and compare quality of life in frail versus non-frail patients. Frailty will be assessed with the CAF score. In a substudy we will analyze the risk of renal insufficiency.

Hypothesis:

Patients deemed frail using the CAF score have increased risk of short-term and long-term complications. With the frailty score in addition to EuroSCORE or STS score, we can better predict complications compared to EuroSCORE or STS score alone.

Method:

A) Patients/study population:

FICS study is a prospective observational study of elderly patients undergoing cardiac surgery at the Department of Cardiothoracic Surgery, Rigshospitalet, Copenhagen University Hospital, Denmark. Expect to include 600 patients during a two years inclusion period. With a minimum of 12 month inclusion period, but all included in the analysis, with a maximum follow-up time.

B) Inclusion criteria:

1. All patients aged above 65 years old
2. Patients referred to elective and subacute cardiac surgery
3. All undergoing CABG (coronary artery bypass grafting), valve replacement and CABG with valve replacement.

C) Exclusions criteria:

1. Emergent surgery
2. Clinically unstable
3. Severe neuropsychiatric impairment
4. No cooperation (psychiatric diagnosis).
5. Reoperations

D) Follow-up:

Patients are followed after discharge by searching The Danish National Registry, which contains informations an all somatic hospital admissions. From which there will be collected a copy of the patient record for all hospital admissions. Patient records will be assessed for pour predefined outcome measures.

Information about vital status will be achieved by searching the Danish Central Civil Register. The cause of death will be obtained from patients records and death certificates.

After 30 days we will contact the patients through phone to ask about their quality of life and intake/changes in medicine and again a follow up in Danish Central Civil Register at 12 month.

E) Substudies:

Study 1, Short-term follow-up:

This study describe the proportion of frail patients in our department undergoing cardiac surgery. We will further compare the number of complications between the two groups.

30-day follow-up comparing frail vs non-frail patients undergoing cardiac surgery:

Primary outcome:

In this study the primary outcome will be 30-day all-cause mortality in frail vs. non-frail patients (hospital mortality or death within 30 days postoperatively).

Secondary outcomes: MACCE (Major Adverse Cardiac and Cerebrovascular Events) including:

* AMI
* Stroke
* Mortality

Tertiary outcomes:

* Stroke
* Renal failure until discharged:
* Prolonged ventilation (>24 h)
* Days in intensive care unit (ICU)
* Readmission in ICU
* Deep sternal wound infection (need for operative intervention and antibiotic therapy, with positive culture)
* Need for reoperation (major bleeding)
* Perioperative complications ex gastrointestinal complication (ischemia, gastric ulcer)
* Days of hospitalization
* Discharged to other hospital or nursing home for ongoing medication or rehabilitation and how many days until discharged to home

Study 2, Long-term follow-up:

This study do a follow up, so the last one included is follow minimum 12 month. And the first one included is followed up until the last is recruited.

12 month follow-up in frail vs non-frail patients undergoing cardiac surgery:

Primary outcome:

In this study the primary outcome is all-cause of mortality after 12 month in frail vs. non-frail patients.

Secondary outcomes: MACCE (Major Adverse Cardiac and Cerebrovascular Events) including:

* AMI:
* Stroke
* Mortality

Tertiary outcomes:

* Discharged to other hospital or nursing home for ongoing medication or rehabilitation and how many days until discharged to home
* Prolonged hospitalization ( > 14 days)
* Number of Re-hospitalization
* New diagnosis and medication ( changes and new)
* Social support (need for more help, both care and tools)
* Other complications.

Study 3,Predicting postoperative Acute Kidney Injury (AKI) in frail vs. non-frail patients undergoing cardiac surgery:

AKS is a major complication after cardiac surgery and associated with increased mortality and morbidity. It has been proven that knowing patients renal reserve before surgery is important, both for predicting mortality and AKI outcomes. Since early detection of these patients may contribute to improving outcomes. Estimation of the renal reserve by Serum creatinine, eGFR, Serum cystatin C, Urinary neutrophil gelatinase-associated lipocalin (NGAL), Cr EDTA Clearance and 24 hr. collection of urine to determine Cr Clearance, protein and albumin. This samples will be collecte on preoperative day, postoperativly day 5 and 3 a follow-up 3 months postoperativley.

Primary outcome: In this study the primary outcome is development of AKI and the severity of AKI in frail vs. non-frail patients, defined as having one of the following:

* Diuresis <0,5ml/kg/hr. for >6 consecutive hours
* Serum creatinine raised by >26umol/L within 48 hours
* serum creatinine rises >1,5 fold from the reference value ( the lowest value recorded within 3 months)

Secondary outcomes:

- Persistent AKI: Having AKI for 48 hours or longer. Study 4, To examine the correlation between frailty score and the other two commonly used surgical risk scores, EuroSCORE and STS and their performance characteristics in patients over the age of 65 undergoing cardiac surgery. This study compare the commonly used risk estimation systems for patients undergoing cardio-surgical procedures, as STS in north America and EuroSCORE in Europe with the frailty score CAF and FORECAST for estimation of mortality and morbidity 30 days and 12 month mortality.

F) The Frailty scoring scale:

CAF:

Evaluation of frailty by using the comprehensive assessment of frailty (CAF) scoring scale of S. Sündermann. [14][15]This is based on a combination of different scoring scales. The first part is based on the Fried criteria: weight loss, self-reported exhaustion, low activity, slowness of gait speed and weakness. Where CAF includes all except weight loss. Self-reported exhaustion are two questions by the original CES-D scale, Center for epidemiological study Depression. Low activity by asking to instrumental activity of daily living (IADL). The IADL used are, walking, housework, outdoor activity, regular sport and others. Following are kilocalories per week calculated by formula: Kilo Cal= (w x frequency of activity x duration of activity)/2. Slowness, speed in meters per second, where the patient walk 4 meters in normal walking speed and weakness through grip strength by pulling as strong as you can the grasp of the dynamometer in kilograms (kg).

The second part is physical performance tests. Testing the balance, how long you can stand still with your feet together, with one feet halfway in front of the other (semi-tandem) and with one feet completely in front of the other one (tandem). At each position the time is measured and put in to frailty table to score points. In the last element of balance the patients is asked to turn around themselves 360 degrees and again the time is obtained. Then testing the body control, get up and down from a chair three times, put on and remove a jacket and pick up a pen from the floor.

The last part is Laboratory tests, including level of serum albumin, Creatinine and calculate Forced expiratory volume in 1 s (FEV1).

At the end two physicians, different from the person observing the CAF test (one cardiac surgeon and one experienced clinician) estimate the patients frailty after the Clinical frailty scale score.

The Clinical frailty scale is from the Canadian Study of Health and Aging, Which is based on a frailty index composed of 70 items, from where you estimate the frailty on a scale 1-7. 1. Very fit: robust, active, energetic, well motivated and fit; these people commonly exercise regularly and are in the most fit group for their age. 2. Well: without active disease, but less fit than people in category 1. 3. Well, with treated comorbid disease: disease symptoms are well controlled compared with those in category 4. 4. Apparently vulnerable: although not frankly dependent, these people commonly complain of being "slowed up" or have disease symptoms. 5. Mildly frail: with limited dependence on others for instrumental activities of daily living. 6. Moderately frail: help is needed with both instrumental and non- instrumental activities of daily living. 7. Severely frail: completely dependent on others for the activities of daily living, or terminally ill.

Finally to get the patients total CAF score, you add each individual test scores together. It has a maximum score of 35 points. That is divided into not frail 1-10, moderately frail 11-25 and severely frail 26-35.

Out from the CAF score, there is a ability to score and use FORECAST (Frailty predicts death One year after elective cardiac surgery test) which include only 5 of CAF items: chair rise, weakness, stair climb, CFS (clinical frailty scale) and Serum creatinine. FORECAST has a maximum score of 14 points, which also is divided into, not frail 0-4, moderately frail 5-7 and severely frail 8-14.[17]

Statistics:

Sample size calculation. Based on the CAF frailty score patients will categorizes into the non-frail group (CAF score <11) or the frail group (CAF score 11 or above). In a previous study Sündermann et al. found that 50% of the patients above 75 years undergoing first time CABG were deemed frail using the CAF score. Furthermore, they observed that 1 year mortality was 7% in the non-frail group versus 14% in frail-group[17] . Based on a power of 80% and a risk of type I error of 5% and the mortality reported above gives an inclusion of at least 300 patients in each group.

Data analysis Categorical data will be presented as numbers and percentages and compared using chi square test or Fischer exact test, as appropriate. Continuous data will be described as means with corresponding standard deviations (SD) and compared using students t-test.

Time to event for the primary and secondary outcomes will be analyzed using a Cox regression model. Survival curves will be illustrated with Kaplan-Meier plots.

A P-value of less than 0.05 will be considered significant.

Administration:

The preoperative testing for frailty will take place in the Department of Cardiothoracic Surgery Rigshospitalet, Copenhagen University Hospital, Denmark.

Economy:

This is a non-profit study. The expenses will be covered by the involving departments at Rigshospitalet. The department of cardiothoracic surgery will cover the costs of a project nurse during the inclusion period.

Ethics:

Today our department use EuroSCORE as a risk score preoperative. The use of frailty score has been used in the department of cardiology the last years.

Admission of frailty scoring in our department is humanly justified since the patient takes no risk and there are no side effects.

We find it financially responsible to introduce, because we hypothetical expect that this will lead to fewer readmissions, fewer ICU days and hospitalization days.

Appendix Definitions Definition MACCE:[18] Non-fatal cardiac arrest: An absence of cardiac rhythm or presence of chaotic rhythm requiring any component of basic or advanced cardiac life support.

Acute myocardial infarction: Increase and gradual decrease in troponin level or a faster increase and decrease of creatine kinase isoenzyme as markers of myocardial necrosis in the company of at least one of the following: ischaemic symptoms, abnormal Q waves on the ECG, ST-segment elevation or depression; or coronary artery intervention (e.g. coronary angioplasty) or a typical decrease in an elevated troponin level detected at its peak after surgery in a patient without a documented alternative explanation for the troponin elevation.

Congestive heart failure: New in-hospital signs or symptoms of dyspnoea or fatigue, orthopnoea, paroxysmal nocturnal dyspnoea, increased jugular venous pressure, pulmonary rales on physical examination, cardiomegaly, or pulmonary vascular engorgement.

New cardiac arrhythmia: ECG evidence of atrial flutter, atrial fibrillation, or second- or third-degree atrioventricular conduction block.

Angina: Dull diffuse substernal chest discomfort precipitated by exertion or emotion and relieved by rest or nitroglycerin.

Stroke: Embolic, thrombotic, or haemorrhagic event lasting at least 30 min with or without persistent residual motor, sensory, or cognitive dysfunction; if the neurological symptoms continue for .24 h, a person is diagnosed with stroke, and if lasting ,24 h the event is defined as a transient ischaemic attack.

Cardiovascular death: Any death, unless an unequivocal non-cardiovascular cause could be established.

Cerebrovascular death: A death caused by cerebrovascular disease.

Renal Failure: diuresis <0,5ml/kg/hr. for >6 consecutive hours or serum creatinine raised by >26umol/L (0,3 mg/dl) within 48 hours or serum creatinine rises >1,5 fold from the reference value at the day 0 to 14.

ELIGIBILITY:
Inclusion Criteria:

* 1) All patients aged above 65 years old 2) Patients referred to elective and subacute cardiac surgery 3) All undergoing CABG (coronary artery bypass grafting), valve replacement and CABG with valve replacement.

Exclusion Criteria:

* Emergency surgery 2) Clinically unstable 3) Severe neuropsychiatric impairment 4) No cooperation (psychiatric diagnosis). 5) Reoperations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We expect to include 600 patients during a two years inclusion period. With a minimum of 12-month follow-up, but all included in the analysis, with maximum follow-up time.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-02; Primary Completion 2018-07 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: In this study the primary outcome will be 30-day all-cause mortality in frail vs non-frail patients (hospital mortality or death within 30 days postoperatively). | 30 days

SECONDARY OUTCOMES:
MACCE (Major Adverse Cardiac and Cerebrovascular Events) including: - AMI: - Stroke - Mortality | 30 days

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldberg RJ, Yarzebski J, Lessard D, Gore JM. A two-decades (1975 to 1995) long experience in the incidence, in-hospital and long-term case-fatality rates of acute myocardial infarction: a community-wide perspective. J Am Coll Cardiol. 1999 May;33(6):1533-9. doi: 10.1016/s0735-1097(99)00040-6. PMID 10334419
- [Background] Alexander KP, Anstrom KJ, Muhlbaier LH, Grosswald RD, Smith PK, Jones RH, Peterson ED. Outcomes of cardiac surgery in patients > or = 80 years: results from the National Cardiovascular Network. J Am Coll Cardiol. 2000 Mar 1;35(3):731-8. doi: 10.1016/s0735-1097(99)00606-3. PMID 10716477
- [Background] Afilalo J, Eisenberg MJ, Morin JF, Bergman H, Monette J, Noiseux N, Perrault LP, Alexander KP, Langlois Y, Dendukuri N, Chamoun P, Kasparian G, Robichaud S, Gharacholou SM, Boivin JF. Gait speed as an incremental predictor of mortality and major morbidity in elderly patients undergoing cardiac surgery. J Am Coll Cardiol. 2010 Nov 9;56(20):1668-76. doi: 10.1016/j.jacc.2010.06.039. PMID 21050978
- [Background] Green P, Woglom AE, Genereux P, Daneault B, Paradis JM, Schnell S, Hawkey M, Maurer MS, Kirtane AJ, Kodali S, Moses JW, Leon MB, Smith CR, Williams M. The impact of frailty status on survival after transcatheter aortic valve replacement in older adults with severe aortic stenosis: a single-center experience. JACC Cardiovasc Interv. 2012 Sep;5(9):974-81. doi: 10.1016/j.jcin.2012.06.011. PMID 22995885
- [Background] Schoenenberger AW, Stortecky S, Neumann S, Moser A, Juni P, Carrel T, Huber C, Gandon M, Bischoff S, Schoenenberger CM, Stuck AE, Windecker S, Wenaweser P. Predictors of functional decline in elderly patients undergoing transcatheter aortic valve implantation (TAVI). Eur Heart J. 2013 Mar;34(9):684-92. doi: 10.1093/eurheartj/ehs304. Epub 2012 Sep 24. PMID 23008508
- [Background] Lee DH, Buth KJ, Martin BJ, Yip AM, Hirsch GM. Frail patients are at increased risk for mortality and prolonged institutional care after cardiac surgery. Circulation. 2010 Mar 2;121(8):973-8. doi: 10.1161/CIRCULATIONAHA.108.841437. Epub 2010 Feb 16. PMID 20159833
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Stortecky S, Schoenenberger AW, Moser A, Kalesan B, Juni P, Carrel T, Bischoff S, Schoenenberger CM, Stuck AE, Windecker S, Wenaweser P. Evaluation of multidimensional geriatric assessment as a predictor of mortality and cardiovascular events after transcatheter aortic valve implantation. JACC Cardiovasc Interv. 2012 May;5(5):489-496. doi: 10.1016/j.jcin.2012.02.012. PMID 22625186
- [Background] Di Dedda U, Pelissero G, Agnelli B, De Vincentiis C, Castelvecchio S, Ranucci M. Accuracy, calibration and clinical performance of the new EuroSCORE II risk stratification system. Eur J Cardiothorac Surg. 2013 Jan;43(1):27-32. doi: 10.1093/ejcts/ezs196. Epub 2012 Jul 20. PMID 22822108
- [Background] Koene BM, van Straten AH, Soliman Hamad MA, Berreklouw E, Ter Woorst JF, Tan ME, van Zundert AJ. Predictive value of the additive and logistic EuroSCOREs in patients undergoing aortic valve replacement. J Cardiothorac Vasc Anesth. 2011 Dec;25(6):1071-5. doi: 10.1053/j.jvca.2011.05.010. Epub 2011 Jul 2. PMID 21723746
- [Background] Qadir I, Salick MM, Perveen S, Sharif H. Mortality from isolated coronary bypass surgery: a comparison of the Society of Thoracic Surgeons and the EuroSCORE risk prediction algorithms. Interact Cardiovasc Thorac Surg. 2012 Mar;14(3):258-62. doi: 10.1093/icvts/ivr072. Epub 2011 Dec 18. PMID 22184465
- [Background] de Arenaza DP, Pepper J, Lees B, Rubinstein F, Nugara F, Roughton M, Jasinski M, Bazzino O, Flather M; ASSERT (Aortic Stentless versus Stented valve assessed by Echocardiography Randomised Trial) Investigators. Preoperative 6-minute walk test adds prognostic information to Euroscore in patients undergoing aortic valve replacement. Heart. 2010 Jan;96(2):113-7. doi: 10.1136/hrt.2008.161174. Epub 2009 Jun 28. PMID 19561363
- [Background] Afilalo J, Mottillo S, Eisenberg MJ, Alexander KP, Noiseux N, Perrault LP, Morin JF, Langlois Y, Ohayon SM, Monette J, Boivin JF, Shahian DM, Bergman H. Addition of frailty and disability to cardiac surgery risk scores identifies elderly patients at high risk of mortality or major morbidity. Circ Cardiovasc Qual Outcomes. 2012 Mar 1;5(2):222-8. doi: 10.1161/CIRCOUTCOMES.111.963157. Epub 2012 Mar 6. PMID 22396586
- [Background] Sundermann SH, Dademasch A, Seifert B, Rodriguez Cetina Biefer H, Emmert MY, Walther T, Jacobs S, Mohr FW, Falk V, Starck CT. Frailty is a predictor of short- and mid-term mortality after elective cardiac surgery independently of age. Interact Cardiovasc Thorac Surg. 2014 May;18(5):580-5. doi: 10.1093/icvts/ivu006. Epub 2014 Feb 3. PMID 24497604
- [Background] Sundermann S, Dademasch A, Praetorius J, Kempfert J, Dewey T, Falk V, Mohr FW, Walther T. Comprehensive assessment of frailty for elderly high-risk patients undergoing cardiac surgery. Eur J Cardiothorac Surg. 2011 Jan;39(1):33-7. doi: 10.1016/j.ejcts.2010.04.013. PMID 20627611
- [Background] Afilalo J, Alexander KP, Mack MJ, Maurer MS, Green P, Allen LA, Popma JJ, Ferrucci L, Forman DE. Frailty assessment in the cardiovascular care of older adults. J Am Coll Cardiol. 2014 Mar 4;63(8):747-62. doi: 10.1016/j.jacc.2013.09.070. Epub 2013 Nov 27. PMID 24291279
- [Background] Sundermann S, Dademasch A, Rastan A, Praetorius J, Rodriguez H, Walther T, Mohr FW, Falk V. One-year follow-up of patients undergoing elective cardiac surgery assessed with the Comprehensive Assessment of Frailty test and its simplified form. Interact Cardiovasc Thorac Surg. 2011 Aug;13(2):119-23; discussion 123. doi: 10.1510/icvts.2010.251884. Epub 2011 Mar 4. PMID 21378017
- [Background] Sabate S, Mases A, Guilera N, Canet J, Castillo J, Orrego C, Sabate A, Fita G, Parramon F, Paniagua P, Rodriguez A, Sabate M; ANESCARDIOCAT Group. Incidence and predictors of major perioperative adverse cardiac and cerebrovascular events in non-cardiac surgery. Br J Anaesth. 2011 Dec;107(6):879-90. doi: 10.1093/bja/aer268. Epub 2011 Sep 2. PMID 21890661
- [Derived] Back C, Hornum M, Jorgensen MB, Lorenzen US, Olsen PS, Moller CH. Comprehensive assessment of frailty score supplements the existing cardiac surgical risk scores. Eur J Cardiothorac Surg. 2021 Sep 11;60(3):710-716. doi: 10.1093/ejcts/ezab127. PMID 33724366
- [Derived] Back C, Hornum M, Jorgensen MB, Lorenzen US, Olsen PS, Moller CH. One-year mortality increases four-fold in frail patients undergoing cardiac surgery. Eur J Cardiothorac Surg. 2021 Jan 4;59(1):192-198. doi: 10.1093/ejcts/ezaa259. PMID 32929483
- [Derived] Back C, Hornum M, Olsen PS, Moller CH. 30-day mortality in frail patients undergoing cardiac surgery: the results of the frailty in cardiac surgery (FICS) copenhagen study. Scand Cardiovasc J. 2019 Dec;53(6):348-354. doi: 10.1080/14017431.2019.1644366. Epub 2019 Jul 23. PMID 31304801